CLINICAL TRIAL: NCT07383532
Title: Effects of Self-Management Education and Follow-Up Telephone Support on Diabetes Self-Management, Treatment Compliance, and Medication Self-Efficacy in Adults With Type 2 Diabetes
Brief Title: Effects of Education and Telephone Support on Type 2 Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Alime Selçuk Tosun, Associate Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/08
Record Dates: First submitted 2026-01-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group or the usual care control group and followed in parallel throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Self-Management Education and Telephone Support (Experimental): Participants in this arm received a structured diabetes self-management education program combined with follow-up telephone support. The intervention consisted of three face-to-face education sessions covering diabetes self-management, treatment compliance, and medication use. In addition, participants received two structured follow-up telephone support calls over a two-month period to reinforce education content, support adherence, and address participant questions. Outcomes were assessed using pre-test and post-test measurements, including diabetes self-management, treatment compliance, medication self-efficacy, and biochemical parameters
  Interventions: Behavioral: Diabetes Self-Management Education and Telephone Support
- Usual Care Control Group (No Intervention): Participants in this arm received usual care for Type 2 diabetes without additional diabetes self-management education or follow-up telephone support. They continued routine clinical follow-up and standard treatment as recommended by healthcare providers. Pre-test and post-test assessments were conducted at the same time points as the intervention group, including measures of diabetes self-management, treatment compliance, medication self-efficacy, and biochemical parameters.

INTERVENTIONS:
Behavioral: Diabetes Self-Management Education and Telephone Support — The intervention consisted of a structured diabetes self-management education program and follow-up telephone support. Participants received three face-to-face education sessions focusing on diabetes self-management, treatment compliance, and medication use. Additionally, two structured follow-up telephone support calls were conducted over a two-month period to reinforce education, support adherence, and address participants' questions.
  Arms: Diabetes Self-Management Education and Telephone Support

SUMMARY:
This study examined the effects of self-management education combined with follow-up telephone support on diabetes self-management, treatment compliance, and medication self-efficacy in adults with Type 2 diabetes. A total of 70 adults with type 2 diabetes were randomly assigned to an intervention group or a control group. Participants in the intervention group received diabetes self-management education and follow-up telephone support while the control group received usual care. Data were collected using the Personal Information Form, the Diabetes Self-Management Scale, the Patient Adherence Scale for Type 2 Diabetes Mellitus Treatment, and the Diabetes Medication Use Self-Efficacy Scale.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of type 2 diabetes for at least 6 months
* Between the ages of 18-64
* Literate
* Planned hospitalisation for at least three days
* Using only insulin or insulin + oral antidiabetics as treatment

Exclusion Criteria:

* Individuals with Type 1
* Gestational diabetes,
* Communication disability
* Psychiatric illness
* Severe complications (retinopathy, neuropathy, nephropathy, diabetic foot, cardiovascular disease)
* Condition that prevents physical activity
* Individuals who could not attend at least two sessions of the diabetes education programme

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Management Scale | Baseline and end of the third month after discharge
  The level of diabetes self-management was assessed using the Diabetes Self-Management Scale. The scale evaluates participants' self-management behaviors across four sub-dimensions: glucose management, diet control, physical activity, and utilization of health services. A minimum score of 0 and a maximum score of 10 is obtained from the total scale and sub-dimensions. Higher scores indicating higher levels of diabetes self-management.

SECONDARY OUTCOMES:
Patient Adherence Scale for Type 2 Diabetes Mellitus Treatment | Baseline and end of the third month after discharge
  Treatment adherence was assessed using the Patient Adherence Scale for Type 2 Diabetes Mellitus Treatment, a validated self-report instrument developed to evaluate adherence behaviors in individuals with Type 2 diabetes. The scale assesses multiple dimensions of attitude and emotional factors, knowledge and personal factors, lifestyle change, feelings of anger, feelings, and behaviours appropriate for adherence, diet bargaining and feelings of denial. The highest score obtained from the scale is 150 and the lowest score is 30. As the score obtained from the scale decreases, the individual's adherence to treatment increases.
Diabetes Medication Use Self-efficacy Scale | Baseline and end of the third month after discharge
  Medication use self-efficacy was assessed using the Diabetes Medication Use Self-Efficacy Scale, a validated instrument measuring individuals' confidence in their ability to use diabetes medications despite potential barriers. The scale evaluates self-efficacy related to obligation, preoccupation, and anxiety associated with medication use. The lowest score in the scale is 19 and the highest score is 57. Higher scores indicate higher levels of medication use self-efficacy.
Glycated hemoglobin | Baseline and end of the third month after discharge
  Glycated hemoglobin (HbA1c) in mmol/mol. This data was obtained from routine blood test results recorded in health records at baseline (during hospital admission) and at the physician follow-up visit three months after discharge.
High-density lipoprotein | Baseline and end of the third month after discharge
  High-density lipoprotein (HDL) in mg/dL. This data was obtained from routine blood test results recorded in health records at baseline (during hospital admission) and at the physician follow-up visit three months after discharge.
Low-density lipoprotein | Baseline and end of the third month after discharge
  Low-density lipoprotein (LDL) in mg/dL. This data was obtained from routine blood test results recorded in health records at baseline (during hospital admission) and at the physician follow-up visit three months after discharge.
Total cholesterol | Baseline and end of the third month after discharge
  Total cholesterol in mg/dL. This data was obtained from routine blood test results recorded in health records at baseline (during hospital admission) and at the physician follow-up visit three months after discharge.
Triglyceride | Baseline and end of the third month after discharge
  Triglyceride in mg/dL. This data was obtained from routine blood test results recorded in health records at baseline (during hospital admission) and at the physician follow-up visit three months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Alime Selçuk Tosun, Assoc. Prof., Principal Investigator — Selcuk University, Faculty of Nursing
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this study will not be shared because the study was conducted solely for internal research purposes, and participant confidentiality and privacy are protected in accordance with institutional ethical approval. Data sharing was not planned in the study protocol.

REFERENCES:
- [Background] Eroglu N, Sabuncu N. The effect of education given to type 2 diabetic individuals on diabetes self-management and self-efficacy: Randomized controlled trial. Prim Care Diabetes. 2021 Jun;15(3):451-458. doi: 10.1016/j.pcd.2021.02.011. Epub 2021 Mar 3. PMID 33674221